CLINICAL TRIAL: NCT03894020
Title: A Study of Disease Progression in Genetically Defined Subjects With Geographic Atrophy (GA) Secondary to Age-related Macular Degeneration (AMD)
Brief Title: GTSCOPE - To Evaluate the Natural Progression of Dry Age-related Macular Degeneration (AMD)
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to the interim analysis demonstrating lack of treatment efficacy.
Sponsor: Gyroscope Therapeutics Limited (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: GTSCOPE; CPPY988A12001 (Other: Novartis)
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Dry Age-related Macular Degeneration; Macular Degeneration; Retinal Disease; Retinal Degeneration; Geographic Atrophy; Macular Atrophy
MeSH Terms: conditions — Macular Degeneration; Retinal Diseases; Retinal Degeneration; Geographic Atrophy; Anetoderma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Samples, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study to evaluate the natural progression of dry AMD in genetically defined subjects

DETAILED DESCRIPTION:
Prospective, observational study to evaluate the natural progression of anatomical and functional visual parameters in genetically defined subjects with GA due to AMD.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with unilateral or bilateral Geographic Atrophy (GA) due to Age-related Macular Degeneration (AMD)
2. BCVA of 40 letters or better using ETDRS charts

Exclusion Criteria:

1. Evidence or history of neovascular Age-related Macular Degeneration (AMD) or diabetic retinopathy
2. Significant ocular or non-ocular disease that would impact the subject's ability to participate in the study
3. Participation in another research study involving an investigational product within the previous 4 weeks or 5 half-lives whichever is longer from the screening/baseline OR received a gene/cell therapy at any time previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Geographic Atrophy (GA) | Up to 96 weeks
  Change from baseline in area of Geographic Atrophy, as assessed by Fundus Auto Fluoresence measured in mm2
Colour Fundus (CF) | Up to 96 weeks
  Change from baseline in Colour Fundus Photography measured in mm2
Retinal Drusen Volume | Up to 96 weeks
  Change from baseline in retinal drusen volume measured in mm3
Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) | Up to 96 weeks
  Change from baseline in ETDRS BCVA reading score
Retinal sensitivity | Up to 96 weeks
  Change from baseline in retinal sensitivity as assessed by microperimetry
Visual Functioning Questionnaire | Up to 96 weeks
  Change from baseline in National Eye Institute Visual Functioning Questionnaire 25-Items Version (NEI VFQ-25) Minimum Score (Best) = 29. Maximum score (Worst) = 149
Medical Events of Interest (MEI) | Up to 96 weeks
  Change from baseline in percentage of Participants with MEI
Monocular and Binocular Reading Performance | Up to 96 weeks
  Change in Monocular and Binocular Reading Performance measured in words/min

CONTACTS AND LOCATIONS:
Locations (71):
- United States (33):
  - Retinal Research Institute (retina consultants of AZ), Phoenix, Arizona
  - Retina Centers PC, Tucson, Arizona
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Byers Eye Institute at Stanford, Palo Alto, California
  - Retina Health Center, Fort Myers, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - University Retina Macula Associates PC, Lemont, Illinois
  - Midwest Eye Institute Northside, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Ophthalamic Consultants of Boston (OCB), Boston, Massachusetts
  - Pepose Vision Institute, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - New Jersey Retina Research Foundation, Vauxhall, New Jersey
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - Columbia University Medical Center, New York, New York
  - Retina Association of Western New York, Rochester, New York
  - Wake Forest Baptist Medical Center - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Casey Eye Institute - OHSU, Portland, Oregon
  - Mid-Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Consultants of Houston-TMC, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research LLC, Willow Park, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Proliance Retina (formally known as Vitreoretinal Associates of Washington), Bellevue, Washington
  - Retina Center Northwest, Silverdale, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
- Australia (2):
  - The University of Melbourne - The Centre for Eye Research Australia (CERA), East Melbourne
  - Lions Eye Institute (LEI) - Nedlands, Nedlands
- France (8):
  - Centre Ophtalmologique Retine Gallien, Bordeaux
  - Centre Hospitalier Intercommunal Creteil, Créteil
  - CHU Dijon - Hôpital Mitterrand, Dijon
  - Hopital de la Croix Rousse - GH Nord, Lyon
  - Centre Paradis Monticelli, Marseille
  - Centre Hospitalier Universitaire de Nantes (CHU de Nantes) - Hotel-Dieu, Nantes
  - Hopital Lariboisiere, Paris
  - Centre Hospitalier Universitaire de Poitiers - Poitiers University Hospital, Poitiers
- Germany (8):
  - EyeNet Baden-Wuerttemberg, Freiburg im Breisgau
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - University Hospital Schleswig-Holstein - Campus Luebeck, Lübeck
  - Klinikum rechts der Isar der Technische Universitaet Muenchen, Munich
  - St. Franziskus-Hospital, Münster
  - MVZ ADTC Siegburg GmbH, Siegburg
  - Augenklinik Sulzbach, Sulzbach
  - Universitaetsklinikum Tuebingen, Tübingen
- Netherlands (2):
  - Amsterdam UMC - Locatie AMC, Amsterdam
  - Radboud Universitair Medisch Centrum, Nijmegen
- Poland (4):
  - Okulistyczna "Jasne Blonia" Sp. z o.o., Lodz, Rojna
  - Specjalistyczny Osrodek Okulistyczny Oculomedica, Bydgoszcz
  - Oftalmika - Prywatna Klinika Okulistyczna, Bydgoszcz
  - Caminomed, Tarnowskie Góry
- Spain (5):
  - Instituto de microcirugía ocular, Barcelona
  - Hospital General de Catalunya Sant Cugat del Valles, Barcelona
  - VISSUM Mirasierra, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
- United Kingdom (9):
  - Burnley General Hospital, Burnley
  - NHS Greater Glasgow and Clyde, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Retina Clinic London, London
  - Manchester Royal Eye Hospital, Manchester
  - John Radcliffe Hospital, Oxford
  - Salisbury NHS Foundation Trust, Salisbury
  - Southampton General Hospital, Southampton
  - Sunderland Eye Infirmary, Sunderland